CLINICAL TRIAL: NCT03616613
Title: Analysis of Aortic Abdominal Aneurysm Prevalence in a Population Pilot Screening Program Based on Primary Care Duplex Ultrasound Evaluation
Brief Title: Aortic Abdominal Aneurysm Pilot Screening Programme
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-AAA-2017-42
Record Dates: First submitted 2018-06-14; First posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Aortic Aneurysm, Abdominal
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Men: Men born in 1952 in Barcelona in health areas depending from Hospital de la Santa Creu i Sant Pau.
  Interventions: Diagnostic Test: ABDOMINAL DUPLEX ULTRASONOGRAPHY
- Women: Aleatory sample of women born in 1952 in Barcelona in health areas depending from Hospital de la Santa Creu i Sant Pau.
  Interventions: Diagnostic Test: ABDOMINAL DUPLEX ULTRASONOGRAPHY

INTERVENTIONS:
Diagnostic Test: ABDOMINAL DUPLEX ULTRASONOGRAPHY — Abdominal ultrasonography performed by both primary care doctors or vascular surgeons in Hospital de la Santa Creu i Sant Pau area

SUMMARY:
Populational abdominal aortic aneurysm (AAA) pilot screening programme performed by duplex ultrasonography in population born in 1952 in health areas depending from Hospital de la Santa Creu i Sant Pau in Barcelona. Descriptive data analysis and cost-effectiveness study will be performed.

DETAILED DESCRIPTION:
Populational abdominal aortic aneurysm (AAA) pilot screening programme performed by duplex ultrasonography in population born in 1952 in areas depending from Hospital de la Santa Creu i Sant Pau in Barcelona. Ultrasonography evaluations will be performed in primary health centers by previously trained doctors according to study protocol and AAA management will be according to United Kingdom's National Health Service screening model. A descriptive analysis will be performed to estimate local population prevalence of AAA in both men and women in order to create the basis for a future state AAA screening programme. A cost-effectiveness analysis will be performed in order to assess optimal screening strategies in our population.

ELIGIBILITY:
Inclusion Criteria:

* All men in our area's population census and an aleatory sample of women born in 1952 living in Hospital de la Santa Creu i Sant Pau area.

Exclusion Criteria:

* Previously detected or operated AAA
* Fragile patients not eligible for AAA repair if needed
* Dead people when contacted
* Eligible people refusing to participate
* Eligible people failed to be contacted twice by our department

Ages: 65 Years to 65 Years | Sex: All
Age Groups: Older Adult
Study Population: All men and a random sample of women born in 1952 in Barcelona in the area that depends from Hospital de la Santa Creu i Sant Pau.
Sampling Method: Probability Sample
Enrollment: 2194 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Abdominal aortic measurement | Days (only one day measurement is performed)
  Ultrasound infrarrenal aortic diameter measurement in mm

SECONDARY OUTCOMES:
Smoking habits | 1 day
  Defined by current smoker, former smoker (more than one year without smoking) or non smoker
Surgical intervention if needed | 1 day
  Registry of kind of intervention and date of intervention
Family AAA history | 1 day
  First or second degree relatives with AAA, or no family AAA history
Personal Cardiovascular Risk Factors | 1 day
  Coronary disease, neurovascular disease, peripheral arterial disease or diabetes mellitus
Dislipidaemia | 1 day
  Altered lipid parameters in blood analysis
Arterial Hypertension | 1 day
  Arterial hypertension under medical treatment
Height | 1 day
  measures in cm
Weight | 1 day
  measures in kg
Abdominal perimeter | 1 day
  measures in cm
Goldberg questionnaire | 1 day
  Complete goldberg anxiety and depression questionnaire. It consists of 12 questions and 5 posible answers for each question, and each answer is rated with 1 to 5 points. Total score above 9 indicates risk of depression.
EuroQOL 5 score | 1 day
  EuroQOL 5 quality of life evaluation questionnaire. It consistis of 5 questions with 3 posible answers for each question, and a visual analogical scale for self health perception. Each combination of answers indicates a pattern of health status that can be rated.

IPD SHARING:
Plan to Share IPD: No